CLINICAL TRIAL: NCT02971137
Title: Pain-related Anxiety Intervention for Smokers With Chronic Pain: A Comparative Effectiveness Trial of Smoking Cessation Counseling for Veterans
Brief Title: Pain and Smoking Study
Acronym: PASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 15-092
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Results first posted 2023-01-04 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Smoking; Pain; Smoking Cessation
Keywords: Smoking; Cigarette Smoking; Veterans; Tobacco Use; Pain
MeSH Terms: conditions — Smoking; Pain; Smoking Cessation; Cigarette Smoking; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smoking Cessation plus CBI (SMK-CBI) (Experimental): An intervention that includes a proactive tele-health intervention combining evidence-based smoking cessation counseling augmented with behavioral approaches for coping with pain
  Interventions: Behavioral: Smoking Cessation plus CBI
- Smoking Cessation Standard (SMK-STD) (Active Comparator): A contact-equivalent control that provides standard smoking cessation telephone counseling
  Interventions: Behavioral: Smoking Cessation Standard

INTERVENTIONS:
Behavioral: Smoking Cessation plus CBI — proactive tele-health intervention combining evidence-based smoking cessation counseling augmented with behavioral approaches for coping with pain
  Other Names: SMK-CBI
  Arms: Smoking Cessation plus CBI (SMK-CBI)
Behavioral: Smoking Cessation Standard — standard telephone-based smoking cessation intervention
  Other Names: SMK-STD
  Arms: Smoking Cessation Standard (SMK-STD)

SUMMARY:
This purpose of this study is to test the telephone delivery of a cognitive behavioral intervention (CBI), for smoking cessation among Veteran smokers with chronic pain

DETAILED DESCRIPTION:
Veterans with chronic pain represent an important population in which to focus smoking cessation efforts. Smoking cessation among patients with chronic medical illnesses substantially decreases morbidity and mortality; yet, many patients (>50%) with chronic pain continue to smoke.

This study aims to test the telephone delivery of a cognitive behavioral intervention (CBI), for smoking cessation among Veteran smokers with chronic pain. Proposed is a randomized comparative effectiveness trial with a two-group design in which 370 Veteran smokers with chronic pain will be randomized to either: 1) smoking cessation plus CBI (SMK-CBI), an intervention that includes a proactive tele-health intervention combining evidence-based smoking cessation counseling augmented with behavioral approaches for coping with pain and a tele-medicine clinic for accessing nicotine replacement therapy (NRT), or 2) smoking cessation telephone counseling control (SMK Control), a contact-equivalent control that provides standard smoking cessation telephone counseling and a tele-medicine clinic for accessing NRT.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled at VA Connecticut or VA Central Western Massachusetts
* Current Cigarette Smokers
* Willing to make quit attempt in next 30 days
* Pain intensity 4 or greater on scale 0-10, self-reported

Exclusion Criteria:

* Non-English speaking
* No access to telephone/Lack of Telephone Access
* Severely impaired hearing
* Active diagnosis
* Terminal Illness
* Refusal to provide informed consent
* Enrolled in concurrent smoking cessation programs/research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Anne Bastian, MD MPH, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Central Western Massachusetts Healthcare System, Leeds, MA, Leeds, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Green KT, Wilson SM, Dennis PA, Runnals JJ, Williams RA, Bastian LA, Beckham JC, Dedert EA, Kudler HS, Straits-Troster K, Gierisch JM, Calhoun PS. Cigarette Smoking and Musculoskeletal Pain Severity Among Male and Female Afghanistan/Iraq Era Veterans. Pain Med. 2017 Sep 1;18(9):1795-1804. doi: 10.1093/pm/pnw339. PMID 28340108
- [Result] Charokopos A, Card ME, Gunderson C, Steffens C, Bastian LA. The Association of Obstructive Sleep Apnea and Pain Outcomes in Adults: A Systematic Review. Pain Med. 2018 Sep 1;19(suppl_1):S69-S75. doi: 10.1093/pm/pny140. PMID 30203008
- [Result] Bastian LA, Driscoll M, DeRycke E, Edmond S, Mattocks K, Goulet J, Kerns RD, Lawless M, Quon C, Selander K, Snow J, Casares J, Lee M, Brandt C, Ditre J, Becker W. Pain and smoking study (PASS): A comparative effectiveness trial of smoking cessation counseling for veterans with chronic pain. Contemp Clin Trials Commun. 2021 Aug 20;23:100839. doi: 10.1016/j.conctc.2021.100839. eCollection 2021 Sep. PMID 34485755
- [Result] Edmond SN, Snow JL, Pomeranz J, Van Cleve R, Black AC, Compton P, Becker WC. Delphi study to explore a new diagnosis for "ineffective" long-term opioid therapy for chronic pain. Pain. 2023 Apr 1;164(4):870-876. doi: 10.1097/j.pain.0000000000002783. Epub 2022 Sep 15. PMID 36448976
- [Derived] Bastian LA, Driscoll MA, Goulet JL, DeRycke EC, Edmond SN, Mattocks KM, Brandt CA, Kravetz J, Akuley SA, Becker WC. Smoking Cessation Among Patients with Chronic Pain in a Comparative Effectiveness Trial. J Gen Intern Med. 2025 Dec 18. doi: 10.1007/s11606-025-10083-x. Online ahead of print. PMID 41413292
- [Derived] Muller RD, Driscoll MA, DeRycke EC, Edmond SN, Becker WC, Bastian LA. Factors associated with participation in a walking intervention for veterans who smoke and have chronic pain. J Behav Med. 2024 Dec;47(6):994-1001. doi: 10.1007/s10865-024-00511-4. Epub 2024 Aug 14. PMID 39143444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Started | 189 | 182
Completed | 145 | 126
Not Completed | 44 | 56
Not completed — Lost to Follow-up | 44 | 56

BASELINE CHARACTERISTICS:
Population: Veteran population who smoked at least 4 cigarettes a week and pain intesity scores >4 for at least 3 months
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD) | Total
Number analyzed (Participants) | 189 | 182 | 371
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 133 | 130 | 263
  >=65 years | 56 | 52 | 108
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 60 [46 to 65] | 60 [53 to 65] | 60 [52 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 26 | 44
  Male | 171 | 156 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 16 | 25
  Not Hispanic or Latino | 179 | 165 | 344
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 50 | 47 | 97
  White | 123 | 112 | 235
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 7 | 14 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 189 | 182 | 371

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Abstained From Smoking Cigarettes at 6months (Prolonged Abstinence)
Description: In the past 6 months, have he/she smoked any in each of 2 consecutive weeks?
Time Frame: 6-month
Population: Veteran population who smoked at least 4 cigarettes a week and pain intensity scores >4 for at least 3 months. There were 227/371 6m responders, non-responders were assumed to continue smoking
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 189 | 182
Participants | 43 | 41

2. Primary Outcome: Number of Participants Who Abstained From Smoking Cigarettes at 12 Months (Prolonged Abstinence)
Description: In the past 6 months, have he/she smoked any in each of 2 consecutive weeks?
Time Frame: 12-month post intervention
Population: Veteran population who smoked at least 4 cigarettes a week and pain intensity scores >4 for at least 3 months. There were 271/371 12m responders, non-responders were assumed to continue smoking
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 189 | 182
Participants | 40 | 38

3. Primary Outcome: Number of Participants Who Abstained From Smoking Part of a Cigarette at 6months (30-day Point Prevalence)
Description: 30-day point prevalence abstinence rates, Have he/she smoked at least part of a cigarette in last 30 days?
Time Frame: 6-month post intervention
Population: There were 227/371 6m responders, no responders were assumed to continue smoking
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 189 | 182
Participants | 23 | 11

4. Primary Outcome: Number of Participants Who Abstained From Smoking Part of a Cigarette at 12 Months (30-day Point Prevalence)
Description: 30-day point prevalence abstinence rates, have he/she smoked at least part of a cigarette in last 30 days?
Time Frame: 12 month post intervention
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 189 | 182
Participants | 25 | 18

5. Secondary Outcome: Change in Brief Pain Inventory (BPI) Pain Intensity, Difference From Baseline to Follow-up at 6 Months
Description: BPI Pain Intensity takes the mean of 4 self-reported numeric rating scale questions about one's pain: worst, least, current, and average pain. Rate pain on a 0 (no pain) to 10 (worst pain imaginable) scale. Veterans will be asked at baseline and after intervention. We are showing the change from baseline to follow-up, a negative score means the pain intensity has decreased.
Time Frame: Baseline to 6-month post intervention
Population: 14 of the 227 6m responders were missing data at least 1Q and were excluded from dataset. All 4Q are needed for BPI pain intensity to be scored.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 110 | 103
score on a scale | -0.7 (1.7) | -0.5 (1.8)

6. Secondary Outcome: Change in Pain Interference, Difference Between Baseline and Follow-up at 6 Months
Description: Pain interference will be measured by the Brief Pain Inventory (BPI). Veterans will be asked at baseline and after intervention. How does pain interfere on a 0 (no interference) to 10 (completely interferes) scale on 7 different facets of living. The total is the mean of all 7 questions. Veterans will be asked at baseline and after intervention. We are showing the change from baseline to follow-up, a negative score means the pain interference has decreased.
Time Frame: Baseline to 6-month post intervention
Population: 20 of the 227 6m responders were missing data at least 4/7Q and were excluded from dataset. At least 50% of questions need to be answered for pain interference to be calculated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 106 | 101
score on a scale | -0.72 (2.4) | -0.36 (2.2)

7. Secondary Outcome: Change in Brief Pain Inventory (BPI) Pain Intensity, Difference in Pain Intensity Between Baseline and 12 Months
Description: as for outcome 5
Time Frame: Baseline to 12-month post-intervention
Population: 24 of the 271 12m responders were missing data at least 1Q and were excluded from dataset. All 4Q are needed for BPI pain intensity to be scored.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 135 | 112
score on a scale | -.044 (1.6) | -0.35 (1.7)

8. Secondary Outcome: Change in Pain Interference, Difference Between Baseline and Interference
Description: as for outcome 6
Time Frame: Baseline to 12-month post intervention
Population: 29 of the 271 12m responders were missing data at least 4/7Q and were excluded from dataset. At least 50% of questions need to be answered for pain interference to be calculated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
Number analyzed (Participants) | 128 | 114
score on a scale | -.56 (2.3) | -.46 (2.1)

ADVERSE EVENTS:
Time Frame: Participants were followed for AE data through duration of their 5 counseling sessions time frame around 3 months.
Arm/Group | Smoking Cessation Plus CBI (SMK-CBI) | Smoking Cessation Standard (SMK-STD)
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/182
Serious Adverse Events (participants affected / at risk) | 0/189 | 0/182
Other Adverse Events (participants affected / at risk) | 0/189 | 0/182

LIMITATIONS AND CAVEATS:
Total enrollment was increased from 370 to 371 due to simultaneous enrollment of last subjects for study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02971137/Prot_SAP_000.pdf